CLINICAL TRIAL: NCT01769898
Title: The Role of Theophylline Plus Low-dose Formoterol-budesonide in Treatment of Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xugang, Medical Doctor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: theophylline in bronchiectasis
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Theophylline; Therapeutic Uses; HDAC; HAT; Random placebo study; ICS(inhaled corticosteroid); corticosteroid; Inhaled corticosteroid
MeSH Terms: conditions — Bronchiectasis | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo+formoterol-budesonide (Placebo Comparator): Placebo(for Theophylline sustained-release tablet) tablet by mouth 100mg every 12hours for 24weeks.
  Inhaled Formoterol-budesonide combined treatment 4.5µg/160µg every 12hours for 24weeks.
  Interventions: Drug: Formoterol-budesonide; Drug: Placebo
- Theophylline+formoterol-budesonide (Experimental): Theophylline sustained-release tablet by mouth 100mg every 12hours for 24weeks.
  Inhaled formoterol-budesonide combined treatment 4.5µg/160µg every 12hours for 24weeks.
  Interventions: Drug: Formoterol-budesonide; Drug: Theophylline

INTERVENTIONS:
Drug: Formoterol-budesonide — Formoterol-budesonide combined treatment (4.5µg/160µg Q12H)
  Other Names: Symbicort tu rbuhaler
Drug: Theophylline — Theophylline 0.1 Q12H
  Other Names: Theophylline Sustained-Release Tablet
  Arms: Theophylline+formoterol-budesonide
Drug: Placebo — Placebo for theophylline 0.1 Q12H
  Arms: Placebo+formoterol-budesonide

SUMMARY:
The purpose of this study is to examine the efficacy and safety of 24 weeks treatment with theophylline plus low-dose formoterol-budesonide in subjects with bronchiectasis.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis is an orphan disease caused by the pathogenic vicious circle including infection, inflammation and airway repair. Today's principle of treatment is to break the cycle of inflammation and infection. Nowadays, most clinical trials are anti-infective treatment by antibiotics trying to break this cycle by reducing the bacterial load, which may cause bacterial resistance. There were still some anti-inflammation trials by using inhaled corticosteroids(ICS). Tsang and Martínez-García showed that inhaled corticosteroids reduced IL-1,IL-8 levels and sputum inflammation cells, and improved sputum volume as well as quality of life, though the corticosteroid must be high dose or medium dose combined with long-acting ß2 adrenergic agonists. As described in asthma and chronic obstructive pulmonary disease(COPD), theophylline can improve the activity of histone deacetylase (HDAC) and then enhanced the anti-inflammatory effect of steroids. We hypothesis that theophylline may have the same effect in subjects with bronchiectasis. Theophylline plus inhaled low-dose formoterol-budesonide may improve quality of life and reduce airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years old with non-cystic fibrosis(CF) bronchiectasis, free from acute exacerbations for at least 3 months.Stable phase of the disease.

Exclusion Criteria:

* Patients with a cigarette smoking history of more than 10 packs-year. Patients with COPD. Patients with traction bronchiectasis due to advanced fibrosis. Patients with known intolerance for theophylline. Patients with asthma. Patients with other disease disturbing outcomes of the trials. Patients without consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life Assessment with St George's Respiratory Questionnaire(SGRQ) and Leicester Cough Questionnaire(LCQ) | Baseline and 24 weeks

SECONDARY OUTCOMES:
Mean number of exacerbations per patient per 24 weeks | Baseline and 24 weeks
  Exacerbations defined by persistent (≥ 24 h) deterioration in at least three respiratory symptoms, including cough, dyspnea, hemoptysis, increased sputum purulence or volume, chest pain (with or without fever).
Changes of sputum characteristics from baseline to 24 weeks | Baseline and 24 weeks
Changes of 24 hour sputum volume from baseline to 24 weeks | Baseline and 24 weeks
Changes of forced expiratory volume in 1 second(FEV1) from baseline to 24 weeks | Baseline and 24 weeks
Changes of mean forced expiratory flow between 25% and 75% of the FVC(FEF25-75)from baseline to 24 weeks | Baseline and 24 weeks
Changes of forced vital capacity(FVC) from baseline to 24 weeks | Baseline and 24 weeks
Changes of peak expiratory flow(PEF) from baseline to 24 weeks | Baseline and 24 weeks
Induced sputum cytology count | Baseline and 24 weeks
Changes of sputum culture from baseline to 24 weeks | Baseline and 24 weeks
IL-6 | Baseline and 24 weeks
  Test IL-6 both in blood and sputum.
IL-8 | Baseline and 24 weeks
  Test IL-8 both in blood and sputum.
IL-10 | At 24 weeks
  Test IL-10 both in blood and sputum.
Tumor necrosis factor(TNF)α | Baseline and 24 weeks
  Test TNF-α both in blood and sputum.
Activity of histone deacetylase(HDAC) | Baseline and 24 weeks
  HDACs are extracted from cells in blood.
Activity of histone acetyltransferase(HAT) | Baseline and 24 weeks
  HATs are extracted from cells in blood.
8-Isoprostane | Baseline and 24 weeks
Neutrophilic granulocytes in blood routine examination | Baseline and 24 weeks
White blood cells in blood routine examination | Baseline and 24 weeks
Monocytes in blood routine examination | Baseline and 24 weeks
Eosinophilic granulocytes in blood routine examination | Baseline and 24 weeks
Number of participants with Adverse events as a measure of safety and tolerability | 24 weeks
  Adverse events may contain symptoms such as nausea, sickness, headache, insomnia, palpitation, arrhythmia and so on. Record the symptoms and times of the patients.
Plasma Concentration of Theophylline | 24 weeks
  Venous blood was taken for plasma theophylline at the end of the treatment period. (At the very time of 2 hours after patients taken the pills)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Rongchang, Professor, Study Director — institute vice director; Zhong Nanshan, Professor, Study Director — institute director
Locations (2):
- China (2):
  - State Key Laboratory of Respiratory Research Institute., Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong